CLINICAL TRIAL: NCT02189018
Title: Activity To Improve Outcomes in Peripheral Arterial Disease
Acronym: ACTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baltimore VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brajesh K Lal, Professor, Baltimore VA Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00059151
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Peripheral Arterial Occlusive Disease
Keywords: Peripheral arterial disease; Endovascular; Exercise; Perfusion; Functional capacity
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1; Peripheral Arterial Disease; Motor Activity | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (Active Comparator): Ad lib activity at home
  Interventions: Other: Ad lib activity at home
- Active Exercise (Experimental): Active exercise on treadmill
  Interventions: Other: Active Exercise
- Neuromuscular electrical stimulation (Experimental): Neuromuscular electrical stimulation
  Interventions: Other: Neuromuscular electrical stimulation
- Weight loss and active exercise (Experimental): Weight loss plus active exercise on treadmill
  Interventions: Other: Weight loss and active exercise

INTERVENTIONS:
Other: Active Exercise — Active exercise on a treadmill
  Arms: Active Exercise
Other: Neuromuscular electrical stimulation — Neuromuscular electrical stimulation
  Arms: Neuromuscular electrical stimulation
Other: Weight loss and active exercise — Weight loss and active exercise on a treadmill
  Arms: Weight loss and active exercise
Other: Ad lib activity at home — Ad lib activity at home
  Arms: Control

SUMMARY:
Peripheral artery disease (PAD) results in blockages of arteries (blood vessels) in the legs and decreased blood flow to the legs. This may cause difficulty or pain with walking or other activities that use leg muscles. Exercise may help improve blood flow in the legs and improve the ability to walk. This research project is being implemented in adults with PAD to examine the effects of exercise or weight loss programs on lower extremity blood flow, health, and physical function.

DETAILED DESCRIPTION:
This pilot study seeks to gather data on different exercise interventions in PAD. Collectively, the proposed studies will gather data on the role of novel exercise interventions in those with PAD who are receiving conservative treatment as well as those who have undergone an endovascular intervention for lower extremity arterial disease.

We hypothesize that patients who undergo an exercise intervention will: A) show improved lower extremity perfusion and B) improve their functional ability, compared to a standard care control group over 6 months of follow-up. We further hypothesize that these improvements are mediated through angiogenesis and increased perfusion of the lower limb, as well as improvements in muscle strength, mass, and function.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-90 years
* Ankle brachial index < 0.9

Exclusion Criteria:

* Cancer under active treatment, except prostate, skin, and hematologic cancers
* Planned for open lower extremity bypass surgery
* Body mass index >45
* Lower extremity gangrene

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Lower extremity perfusion | 6 months
  Ankle brachial index and ultrasound quantification of muscle perfusion

SECONDARY OUTCOMES:
Functional capacity | 6 months
  Treadmill exercise testing

CONTACTS AND LOCATIONS:
Overall Officials: Brajesh K Lal, MD, Principal Investigator — Baltimore VAMC, University of Maryland School of Medicine
Locations (1):
- Baltimore VAMC, Baltimore, Maryland, United States